CLINICAL TRIAL: NCT03055247
Title: A Multicentric, Exploratory, Non-randomised, Non-controlled, Prospective, Open-label Phase II Study Evaluating Safety and Efficacy of IBU, G-CSF and Plerixafor as Stem Cell Mobilization Regimen in Patients Affected by X-CGD
Brief Title: Combination of Ibuprofen, G-CSF and Plerixafor as Stem Cells Mobilization Regimen in Patients Affected by X-CGD
Acronym: XCGD-MOBI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Fondazione Telethon (Other)
Responsible Party: Principal Investigator, Ciceri Fabio, Director Hematology and BMT Unit, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-002356-27
Record Dates: First submitted 2016-07-21; First posted 2017-02-16 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Chronic Granulomatous Disease X-linked (X-CGD)
Keywords: Chronic granulomatous disease X-linked; Ibuprofen; Mobilization regimen; Gene Therapy
MeSH Terms: conditions — Granulomatous Disease, Chronic | interventions — Ibuprofen; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XCGD mobilization (Experimental): Treatment with combination of Ibuprofen, Myelostim and Mozobil
  Interventions: Drug: Ibuprofen; Drug: Myelostim; Drug: Mozobil

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen: 3 mg/kg tid (total daily dose: 9 mg/kg); administered orally from day 1 to day 5 and then from day 14 to the day before the last LP.
Drug: Myelostim — Myelostim (G-CSF): 5 µg/kg bid (total daily dose 10 µg/kg); administered subcutaneously from day 19 to the day of the last LP.
Drug: Mozobil — Mozobil (Plerixafor): 0,24 mg/kg daily. When CD34+ are ≥ 10 /μL Plerixafor will be administered subcutaneously from the next day (or from day 24 if CD34+ are < 10 /μL) to the day of the last LP.

SUMMARY:
This is a phase II exploratory study conducted to evaluate the safety and efficacy of the combination of Ibuprofen, G-CSF and Plerixafor as stem cell mobilization regimen in patients affected by X-CGD.

DETAILED DESCRIPTION:
We designed a mobilization trial with the aim of collecting a sufficient number of HSPC in X-CGD patients; it is well known that this procedure is challenging for these patients, potentially due to functional defects induced by their chronic inflammatory state.

The combination of G-CSF and Plerixafor is considered state of the art for HSPC harvest in gene therapy trials; we considered to add a non-steroidal inflammatory drug to increase HSPC mobilization and reduce inflammation that could have a role in altering HSPC content.

If this trial confirms the synergistic effect of the three drugs under investigation, such a regimen will be considered for a HSPC mobilization in future gene therapy trial for X-CGD patients.

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of X-CGD
* 18-45 years of age
* Karnofsky Index > 80 %
* Adequate cardiac, renal, hepatic and pulmonary function.
* Negative thrombophilic screen and negative history for previous thrombotic events
* Written informed consent

Exclusion Criteria:

* Previous Bone Marrow Transplantation or previous Gene Therapy.
* Use of other investigational agents within 4 weeks prior to study enrolment (within 6 weeks if use of long-acting agents).
* Ongoing IFN-γ treatment (within 4 weeks).
* Symptomatic inflammatory bowel disease.
* Symptomatic viral, bacterial, or fungal infection within 6 weeks of eligibility
* Neoplasia (except local skin cancer) or history of "familial" cancer
* Myelodysplasia or other serious hematological disorder
* History of uncontrolled seizures and deep venous thrombosis
* Other systemic disease judged as incompatible with the procedure
* Positivity for HIV and/or HCV RNA and/or HbsAg and/or HBV DNA
* Active alcohol or substance abuse within 6 months of the study.
* Contraindications to IBU, G-CSF, Plerixafor or Pantoprazole administration

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2015-11-06 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2026-07-18 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients experiencing adverse events | up to 30 days after the last LP
  Percentage of patients experiencing adverse events, as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse events (CTCAe v3.0, 2006) (all grades).
Number of CD34+ collected per body weight after the last LP | Day 21-24
  Cytofluorimetric analysis for CD34 on PB and on collected PBSC to calculate the number of CD34+ cells collected per kg body weight. The analysis will be performed at the end of the LP(s) (Day 21-24)

SECONDARY OUTCOMES:
Change in number of CD34+ cells in PB before and after administration of Ibuprofen | Day 6 and day 7
  Cytofluorimetric analysis to determine the number of CD34+ cells present in PB on day 6 and 7 compared to before the administration of Ibuprofen
Transduction efficiency | Through study completion, an average of 1 year
  Efficient transduction of mobilized HSPC with a lentiviral vector encoding for a corrective cDNA of the human gp91phox gene. Frequency and Vector Copy Number tested by PCR.
DHR (dihydrorhodamine) test in myeloid progeny | Through study completion, an average of 1 year
  Correction of the functional defects in the differentiated myeloid progeny
Functional characterization of mobilized CD34+ cells. | Through study completion, an average of 1 year
  Phenotype analysis (FACS).
Functional characterization of mobilized CD34+ cells. | Through study completion, an average of 1 year
  Clonogenic activity (CFU-C) before and after transduction.
Functional characterization of mobilized CD34+ cells. | Through study completion, an average of 1 year
  Repopulating activity of mobilized CD34+ cells in immunodeficient mice.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Ciceri, MD, PhD, Principal Investigator — Ospedale San Raffaele; Franco Locatelli, MD, PhD, Principal Investigator — Ospedale Pediatrico Bambino Gesù
Locations (2):
- Italy (2):
  - Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - Ospedale San Raffaele, Milan, Lombardy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aiuti A, Bacchetta R, Seger R, Villa A, Cavazzana-Calvo M. Gene therapy for primary immunodeficiencies: Part 2. Curr Opin Immunol. 2012 Oct;24(5):585-91. doi: 10.1016/j.coi.2012.07.012. Epub 2012 Aug 18. PMID 22909900
- [Background] Chiriaco M, Farinelli G, Capo V, Zonari E, Scaramuzza S, Di Matteo G, Sergi LS, Migliavacca M, Hernandez RJ, Bombelli F, Giorda E, Kajaste-Rudnitski A, Trono D, Grez M, Rossi P, Finocchi A, Naldini L, Gentner B, Aiuti A. Dual-regulated lentiviral vector for gene therapy of X-linked chronic granulomatosis. Mol Ther. 2014 Aug;22(8):1472-1483. doi: 10.1038/mt.2014.87. Epub 2014 May 29. PMID 24869932
- [Background] Di Matteo G, Giordani L, Finocchi A, Ventura A, Chiriaco M, Blancato J, Sinibaldi C, Plebani A, Soresina A, Pignata C, Dellepiane RM, Trizzino A, Cossu F, Rondelli R, Rossi P, De Mattia D, Martire B; IPINET (Italian Network for Primary Immunodeficiencies). Molecular characterization of a large cohort of patients with Chronic Granulomatous Disease and identification of novel CYBB mutations: an Italian multicenter study. Mol Immunol. 2009 Jun;46(10):1935-41. doi: 10.1016/j.molimm.2009.03.016. Epub 2009 May 1. PMID 19410294
- [Background] Edmonson JH, Hartmann LC, Long HJ, Colon-Otero G, Fitch TR, Jefferies JA, Braich TA, Maples WJ. Granulocyte-macrophage colony-stimulating factor. Preliminary observations on the influences of dose, schedule, and route of administration in patients receiving cyclophosphamide and carboplatin. Cancer. 1992 Nov 15;70(10):2529-39. doi: 10.1002/1097-0142(19921115)70:103.0.co;2-h. PMID 1423182
- [Background] Gennery AR, Slatter MA, Grandin L, Taupin P, Cant AJ, Veys P, Amrolia PJ, Gaspar HB, Davies EG, Friedrich W, Hoenig M, Notarangelo LD, Mazzolari E, Porta F, Bredius RG, Lankester AC, Wulffraat NM, Seger R, Gungor T, Fasth A, Sedlacek P, Neven B, Blanche S, Fischer A, Cavazzana-Calvo M, Landais P; Inborn Errors Working Party of the European Group for Blood and Marrow Transplantation; European Society for Immunodeficiency. Transplantation of hematopoietic stem cells and long-term survival for primary immunodeficiencies in Europe: entering a new century, do we do better? J Allergy Clin Immunol. 2010 Sep;126(3):602-10.e1-11. doi: 10.1016/j.jaci.2010.06.015. Epub 2010 Jul 31. PMID 20673987
- [Background] Grez M, Reichenbach J, Schwable J, Seger R, Dinauer MC, Thrasher AJ. Gene therapy of chronic granulomatous disease: the engraftment dilemma. Mol Ther. 2011 Jan;19(1):28-35. doi: 10.1038/mt.2010.232. Epub 2010 Nov 2. PMID 21045810
- [Background] Gungor T, Teira P, Slatter M, Stussi G, Stepensky P, Moshous D, Vermont C, Ahmad I, Shaw PJ, Telles da Cunha JM, Schlegel PG, Hough R, Fasth A, Kentouche K, Gruhn B, Fernandes JF, Lachance S, Bredius R, Resnick IB, Belohradsky BH, Gennery A, Fischer A, Gaspar HB, Schanz U, Seger R, Rentsch K, Veys P, Haddad E, Albert MH, Hassan M; Inborn Errors Working Party of the European Society for Blood and Marrow Transplantation. Reduced-intensity conditioning and HLA-matched haemopoietic stem-cell transplantation in patients with chronic granulomatous disease: a prospective multicentre study. Lancet. 2014 Feb 1;383(9915):436-48. doi: 10.1016/S0140-6736(13)62069-3. Epub 2013 Oct 23. PMID 24161820
- [Background] Holland SM. Chronic granulomatous disease. Clin Rev Allergy Immunol. 2010 Feb;38(1):3-10. doi: 10.1007/s12016-009-8136-z. PMID 19504359
- [Background] Hong KT, Kang HJ, Kim NH, Kim MS, Lee JW, Kim H, Park KD, Shin HY, Ahn HS. Successful mobilization using a combination of plerixafor and G-CSF in pediatric patients who failed previous chemomobilization with G-CSF alone and possible complications of the treatment. J Hematol Oncol. 2012 Mar 30;5:14. doi: 10.1186/1756-8722-5-14. PMID 22458355
- [Background] Hoggatt J, Mohammad KS, Singh P, Hoggatt AF, Chitteti BR, Speth JM, Hu P, Poteat BA, Stilger KN, Ferraro F, Silberstein L, Wong FK, Farag SS, Czader M, Milne GL, Breyer RM, Serezani CH, Scadden DT, Guise TA, Srour EF, Pelus LM. Differential stem- and progenitor-cell trafficking by prostaglandin E2. Nature. 2013 Mar 21;495(7441):365-9. doi: 10.1038/nature11929. Epub 2013 Mar 13. PMID 23485965
- [Background] Kang EM, Choi U, Theobald N, Linton G, Long Priel DA, Kuhns D, Malech HL. Retrovirus gene therapy for X-linked chronic granulomatous disease can achieve stable long-term correction of oxidase activity in peripheral blood neutrophils. Blood. 2010 Jan 28;115(4):783-91. doi: 10.1182/blood-2009-05-222760. Epub 2009 Dec 1. PMID 19965657
- [Background] Kang HJ, Bartholomae CC, Paruzynski A, Arens A, Kim S, Yu SS, Hong Y, Joo CW, Yoon NK, Rhim JW, Kim JG, Von Kalle C, Schmidt M, Kim S, Ahn HS. Retroviral gene therapy for X-linked chronic granulomatous disease: results from phase I/II trial. Mol Ther. 2011 Nov;19(11):2092-101. doi: 10.1038/mt.2011.166. Epub 2011 Aug 30. PMID 21878903
- [Background] Martinez CA, Shah S, Shearer WT, Rosenblatt HM, Paul ME, Chinen J, Leung KS, Kennedy-Nasser A, Brenner MK, Heslop HE, Liu H, Wu MF, Hanson IC, Krance RA. Excellent survival after sibling or unrelated donor stem cell transplantation for chronic granulomatous disease. J Allergy Clin Immunol. 2012 Jan;129(1):176-83. doi: 10.1016/j.jaci.2011.10.005. Epub 2011 Nov 12. PMID 22078471
- [Background] Ott MG, Schmidt M, Schwarzwaelder K, Stein S, Siler U, Koehl U, Glimm H, Kuhlcke K, Schilz A, Kunkel H, Naundorf S, Brinkmann A, Deichmann A, Fischer M, Ball C, Pilz I, Dunbar C, Du Y, Jenkins NA, Copeland NG, Luthi U, Hassan M, Thrasher AJ, Hoelzer D, von Kalle C, Seger R, Grez M. Correction of X-linked chronic granulomatous disease by gene therapy, augmented by insertional activation of MDS1-EVI1, PRDM16 or SETBP1. Nat Med. 2006 Apr;12(4):401-9. doi: 10.1038/nm1393. Epub 2006 Apr 2. PMID 16582916
- [Background] Panch SR, Yau YY, Kang EM, De Ravin SS, Malech HL, Leitman SF. Mobilization characteristics and strategies to improve hematopoietic progenitor cell mobilization and collection in patients with chronic granulomatous disease and severe combined immunodeficiency. Transfusion. 2015 Feb;55(2):265-74. doi: 10.1111/trf.12830. Epub 2014 Aug 21. PMID 25143186
- [Background] Pham HP, Patel N, Semedei-Pomales M, Bhatia M, Schwartz J. The use of plerixafor in hematopoietic progenitor cell collection in pediatric patients: a single center experience. Cytotherapy. 2012 Apr;14(4):467-72. doi: 10.3109/14653249.2012.658912. Epub 2012 Feb 20. PMID 22339604
- [Background] Roos D, Kuhns DB, Maddalena A, Bustamante J, Kannengiesser C, de Boer M, van Leeuwen K, Koker MY, Wolach B, Roesler J, Malech HL, Holland SM, Gallin JI, Stasia MJ. Hematologically important mutations: the autosomal recessive forms of chronic granulomatous disease (second update). Blood Cells Mol Dis. 2010 Apr 15;44(4):291-9. doi: 10.1016/j.bcmd.2010.01.009. Epub 2010 Feb 18. PMID 20167518
- [Background] Sevilla J, Schiavello E, Madero L, Pardeo M, Guggiari E, Baragano M, Luksch R, Massimino M. Priming of hematopoietic progenitor cells by plerixafor and filgrastim in children with previous failure of mobilization with chemotherapy and/or cytokine treatment. J Pediatr Hematol Oncol. 2012 Mar;34(2):146-50. doi: 10.1097/MPH.0b013e31821c2cb8. PMID 22009006
- [Background] Seger RA. Modern management of chronic granulomatous disease. Br J Haematol. 2008 Feb;140(3):255-66. doi: 10.1111/j.1365-2141.2007.06880.x. PMID 18217895
- [Background] Santilli G, Almarza E, Brendel C, Choi U, Beilin C, Blundell MP, Haria S, Parsley KL, Kinnon C, Malech HL, Bueren JA, Grez M, Thrasher AJ. Biochemical correction of X-CGD by a novel chimeric promoter regulating high levels of transgene expression in myeloid cells. Mol Ther. 2011 Jan;19(1):122-32. doi: 10.1038/mt.2010.226. Epub 2010 Oct 26. PMID 20978475
- [Background] Seger RA. Chronic granulomatous disease: recent advances in pathophysiology and treatment. Neth J Med. 2010 Nov;68(11):334-40. PMID 21116026
- [Background] Son MH, Kang ES, Kim DH, Lee SH, Yoo KH, Sung KW, Koo HH, Kim DW, Kim JY, Cho EJ. Efficacy and toxicity of plerixafor for peripheral blood stem cell mobilization in children with high-risk neuroblastoma. Pediatr Blood Cancer. 2013 Aug;60(8):E57-9. doi: 10.1002/pbc.24506. Epub 2013 Mar 4. PMID 23460590
- [Background] Stein S, Ott MG, Schultze-Strasser S, Jauch A, Burwinkel B, Kinner A, Schmidt M, Kramer A, Schwable J, Glimm H, Koehl U, Preiss C, Ball C, Martin H, Gohring G, Schwarzwaelder K, Hofmann WK, Karakaya K, Tchatchou S, Yang R, Reinecke P, Kuhlcke K, Schlegelberger B, Thrasher AJ, Hoelzer D, Seger R, von Kalle C, Grez M. Genomic instability and myelodysplasia with monosomy 7 consequent to EVI1 activation after gene therapy for chronic granulomatous disease. Nat Med. 2010 Feb;16(2):198-204. doi: 10.1038/nm.2088. Epub 2010 Jan 24. PMID 20098431
- [Background] Yannaki E, Karponi G, Zervou F, Constantinou V, Bouinta A, Tachynopoulou V, Kotta K, Jonlin E, Papayannopoulou T, Anagnostopoulos A, Stamatoyannopoulos G. Hematopoietic stem cell mobilization for gene therapy: superior mobilization by the combination of granulocyte-colony stimulating factor plus plerixafor in patients with beta-thalassemia major. Hum Gene Ther. 2013 Oct;24(10):852-60. doi: 10.1089/hum.2013.163. PMID 24001178
- [Background] Yannaki E, Papayannopoulou T, Jonlin E, Zervou F, Karponi G, Xagorari A, Becker P, Psatha N, Batsis I, Kaloyannidis P, Tahynopoulou V, Constantinou V, Bouinta A, Kotta K, Athanassiadou A, Anagnostopoulos A, Fassas A, Stamatoyannopoulos G. Hematopoietic stem cell mobilization for gene therapy of adult patients with severe beta-thalassemia: results of clinical trials using G-CSF or plerixafor in splenectomized and nonsplenectomized subjects. Mol Ther. 2012 Jan;20(1):230-8. doi: 10.1038/mt.2011.195. Epub 2011 Sep 27. PMID 21952171
- [Background] Wu C, Dunbar CE. Stem cell gene therapy: the risks of insertional mutagenesis and approaches to minimize genotoxicity. Front Med. 2011 Dec;5(4):356-71. doi: 10.1007/s11684-011-0159-1. Epub 2011 Dec 27. PMID 22198747